CLINICAL TRIAL: NCT04399421
Title: Pedicle Screw Fixation in Osteoporotic Patients With Degenerative Lumbar Diseases: a Prospective Cohort Study
Brief Title: Pedicle Screw Fixation in Osteoporotic Lumbar Spine
Acronym: PSFOLS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BYSYDL2019006
Record Dates: First submitted 2020-05-19; First posted 2020-05-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Osteoporosis; Degenerative Lumbar Diseases
Keywords: Osteoporosis; Pedicle screw fixation; Degenerative lumbar diseases
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional pedicle screw fixation: Patients undergoing conventional pedicle screw fixation without the use of bone cement.
- Cement-augmented pedicle screw fixation: Patients undergoing pedicle screw fixation augmented with bone cement.

SUMMARY:
This is a prospective, observational single-center study. The osteoporotic patients requiring pedicle screw fixation for lumbar degenerative diseases are prospectively enrolled and followed up. This study mainly focuses on the most common osteoporosis-related surgical complications, which are pedicle screw loosening and the failure of lumbar fusion. The global and local bone mineral density(BMD) are evaluated with DXA, vertebral CT Hounsfield units(HU) before the surgery. The mechanical strength of the bone mass within the screw trajectory is also measured with a customized device during the surgery. We explored the effect of BMD on the pedicle screw loosening rate and fusion rate. In addition, the patients undergoing lumbar fixation with conventional pedicle screws without the use of bone cement are compared with those undergoing the fixation augmented with bone cement. The objective is to offer more detailed clinical evidence to guide the use of pedicle screw augmentation techniques in osteoporotic patients.

DETAILED DESCRIPTION:
Pedicle screw fixation is a widely used technique for the surgical treatment of degenerative lumbar diseases, which can stabilize the spine before solid fusion and restore spinal balance. However, because of population aging and the high rate of osteoporosis in the elderly with lumbar degenerative diseases, the pedicle screw loosening has become a frequently reported complication. The bone-screw interface in osteoporotic spine is unstable, leading to reduced pull-out force and cut-out force.

Previous studies have widely reported the bone cement augmentation techniques used to directly strengthen the pedicle screws. It has been proved that cement-augmented pedicle screw fixation is associated with lower loosening rate and higher fusion rate. However, the use of cement can lead to cement leakage and pulmonary embolism, and need extra cost. Therefore, it is very important to identify the correlation between degree of osteoporosis and screw loosening risk , and to establish the indications for cement augmentation in osteoporotic patients.

The osteoporotic patients requiring posterior lumbar fusion with pedicle screw fixation are prospectively enrolled and followed up. The researchers will invite appropriate patients to participate in the study after their surgical plans are determined. General patients data are collected after informed consent, such as age, gender, weight, height, bone mineral density measured in T-scores and Hounsfield units, the mechanical strength of the bone mass within the screw trajectory, detailed surgical plans, and etc. They are followed up at 3, 6, 12, and 24 months according to our clinical routine, including lumbar x-ray and certain questions about the clinical outcomes. In addition, this study requires the patients to have lumbar CT scans because its advantage in judging the fusion status. In addition, the ODI and VAS scores are also routinely recorded.

The patients undergoing conventional pedicle screw fixation without cement augmentation are compared with those undergoing the fixation augmented with bone cement. The primary endpoints are the loosening rate and fusion rate at 12 months follow-up. The secondary endpoints are the loosening rate and fusion rate at other time point of follow-up , and the clinical outcomes(ODI and VAS) at every follow-up. We also explored the correlation between the BMD information measured with different methods and the patients outcomes, in order to find the high-risk patient group.

ELIGIBILITY:
Inclusion Criteria:

* aged≥ 50 years old
* lumbar degenerative diseases requiring lumbar fusion with pedicle screw fixation, such as degenerative lumbar spinal stenosis, degenerative lumbar spondylolisthesis and etc.
* no response to nonoperative treatment of at least 3 months
* osteoporosis diagnosed by any method for bone mineral density evaluation, such as DXA, QCT, or vertebral Hounsfield units
* informed consent

Exclusion Criteria:

* no lumbar CT scans within 3 months before the surgery
* no dual energy x-ray absorptiometry within 6 months before the surgery
* history of lumbar fusion surgery
* cervical myelopathy, thoracic spinal stenosis, motor neuron disease, tuberculosis of spine, spinal tumor

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the orthopaedic department of the Peking University Third Hospital, the osteoporotic in-patients requiring lumbar pedicle screw fixation for lumbar degenerative diseases are invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pedicle screw loosening | 12 months
  The presence of radiolucent zones of ≥1mm thick around any pedicle screw, broken screws, or obvious screw back-out and cut-out on x-ray or CT images
Lumbar fusion | 12 months
  The presence of continuous fusion mass at any fusion segment in CT scans and no obvious intervertebral mobility at any fusion segment on lateral flexion-extension x-ray images.

SECONDARY OUTCOMES:
Pedicle screw loosening | 3 months; 6 months; 24 months
  The presence of radiolucent zones of ≥1mm thick around any pedicle screw, broken screws, or obvious screw back-out and cut-out on x-ray or CT images
Lumbar fusion | 3 months; 6 months; 24 months
  The presence of continuous fusion mass at any fusion segment in CT scans and no obvious intervertebral mobility at any fusion segment on lateral flexion-extension x-ray images.
The Oswestry Disability Index（ODI） | 3 months; 12 months; 6 months; 24 months
  The Oswestry Disability Index (ODI) (%，0-100) is used to assess disability.
VAS score for low back pain | 3 months; 12 months; 6 months; 24 months
  The Visual Analog Scale (VAS 0-10) is used the evaluate low back pain.
VAS score for leg pain | 3 months; 12 months; 6 months; 24 months
  The Visual Analog Scale (VAS 0-10) is used the evaluate leg pain.

CONTACTS AND LOCATIONS:
Overall Officials: Weishi Li, M.D., Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
We will make the clinical study report available half a year after the publication of the results of the study.
Supporting Information: CSR
Time Frame: The IPD will become available half a year after the publication of the results of the study.

REFERENCES:
- [Background] Pannell WC, Savin DD, Scott TP, Wang JC, Daubs MD. Trends in the surgical treatment of lumbar spine disease in the United States. Spine J. 2015 Aug 1;15(8):1719-27. doi: 10.1016/j.spinee.2013.10.014. Epub 2013 Oct 31. PMID 24184652
- [Background] Amirouche F, Solitro GF, Magnan BP. Stability and Spine Pedicle Screws Fixation Strength-A Comparative Study of Bone Density and Insertion Angle. Spine Deform. 2016 Jul;4(4):261-267. doi: 10.1016/j.jspd.2015.12.008. Epub 2016 Jun 16. PMID 27927514
- [Background] Okuyama K, Abe E, Suzuki T, Tamura Y, Chiba M, Sato K. Influence of bone mineral density on pedicle screw fixation: a study of pedicle screw fixation augmenting posterior lumbar interbody fusion in elderly patients. Spine J. 2001 Nov-Dec;1(6):402-7. doi: 10.1016/s1529-9430(01)00078-x. PMID 14588296
- [Background] Bredow J, Boese CK, Werner CM, Siewe J, Lohrer L, Zarghooni K, Eysel P, Scheyerer MJ. Predictive validity of preoperative CT scans and the risk of pedicle screw loosening in spinal surgery. Arch Orthop Trauma Surg. 2016 Aug;136(8):1063-7. doi: 10.1007/s00402-016-2487-8. Epub 2016 Jun 16. PMID 27312862
- [Background] Galbusera F, Volkheimer D, Reitmaier S, Berger-Roscher N, Kienle A, Wilke HJ. Pedicle screw loosening: a clinically relevant complication? Eur Spine J. 2015 May;24(5):1005-16. doi: 10.1007/s00586-015-3768-6. Epub 2015 Jan 24. PMID 25616349
- [Background] Tokuhashi Y, Matsuzaki H, Oda H, Uei H. Clinical course and significance of the clear zone around the pedicle screws in the lumbar degenerative disease. Spine (Phila Pa 1976). 2008 Apr 15;33(8):903-8. doi: 10.1097/BRS.0b013e31816b1eff. PMID 18404111
- [Background] Goldstein CL, Brodke DS, Choma TJ. Surgical Management of Spinal Conditions in the Elderly Osteoporotic Spine. Neurosurgery. 2015 Oct;77 Suppl 4:S98-107. doi: 10.1227/NEU.0000000000000948. PMID 26378363
- [Background] Janssen I, Ryang YM, Gempt J, Bette S, Gerhardt J, Kirschke JS, Meyer B. Risk of cement leakage and pulmonary embolism by bone cement-augmented pedicle screw fixation of the thoracolumbar spine. Spine J. 2017 Jun;17(6):837-844. doi: 10.1016/j.spinee.2017.01.009. Epub 2017 Jan 17. PMID 28108403
- [Background] Zou D, Muheremu A, Sun Z, Zhong W, Jiang S, Li W. Computed tomography Hounsfield unit-based prediction of pedicle screw loosening after surgery for degenerative lumbar spine disease. J Neurosurg Spine. 2020 Jan 3;32(5):716-721. doi: 10.3171/2019.11.SPINE19868. Print 2020 May 1. PMID 31899883
- [Background] Zou D, Jiang S, Zhou S, Sun Z, Zhong W, Du G, Li W. Prevalence of Osteoporosis in Patients Undergoing Lumbar Fusion for Lumbar Degenerative Diseases: A Combination of DXA and Hounsfield Units. Spine (Phila Pa 1976). 2020 Apr 1;45(7):E406-E410. doi: 10.1097/BRS.0000000000003284. PMID 31725127
- [Background] Zou D, Li W, Deng C, Du G, Xu N. The use of CT Hounsfield unit values to identify the undiagnosed spinal osteoporosis in patients with lumbar degenerative diseases. Eur Spine J. 2019 Aug;28(8):1758-1766. doi: 10.1007/s00586-018-5776-9. Epub 2018 Oct 10. PMID 30306332